CLINICAL TRIAL: NCT03932383
Title: 3-D Printer Custom Modified Continuous Positive Airway Pressure Masks to Improve Efficacy and Patient Compliance in Obstructive Sleep Apnea Management
Brief Title: 3D Printer Modified CPAP Mask for Obstructive Sleep Apnea
Acronym: 3DCPAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000100
Record Dates: First submitted 2019-02-21; First posted 2019-04-30 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Cohort study of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Modified CPAP (Experimental): Single arm cohort study of modified mask
  Interventions: Device: Custom CPAP mask

INTERVENTIONS:
Device: Custom CPAP mask — Modified CPAP mask based on 3D image capture

SUMMARY:
This is a prospective pilot to investigate the effect of 3D printer customized CPAP masks on the comfort of patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
Purpose:

The purpose of this protocol is to perform a prospective pilot clinical study to customize patient CPAP masks to reduce air leak in patients with obstructive sleep apnea (OSA). Using 3-D printer-based technology modeling of patient facial features, patient FDA-approved CPAP masks will be modified by strategically applying silicone pads on the CPAP mask to mold to the specific facial features to optimize the CPAP mask-patient interface, improve CPAP mask fit and comfort, reduce air leak, limit air pressure loss and improve compliance with CPAP treatment strategy (as measured over a 30 day trial period).

Protocol:

Potential subjects for this study will be identified at the outpatient Sleep Disorders Clinic at BIDMC. Patients will have documented OSA, prescribed CPAP as standard-of-care, and demonstrate consistent problems with CPAP mask-patient interface with documented high air loss, and poor adherence/ compliance. All potential subjects will have used and will continue to use an FDA-approved CPAP mask selected by the patient.

Potential subjects (along with their FDA-approved CPAP mask) will then be referred to the BIDMC Specialties Clinic and screened, including review of the medical history of OSA, review of documented reports of excessive air leak and suboptimal adherence to CPAP, brief physical exam (esp. focusing on the head-and-neck exam) including assessment of the CPAP mask-patient interface, review of the purpose and goals of the pilot clinical study, a dynamic video of the study subject face will be performed, video downloaded to a computer which will then be used to generate a 3-dimensional plastic model of the study subject face using state-of-the-art 3D printer technology (see details below). The patient's FDA-approved CPAP mask will then be applied to his plastic model of the study subject face, and the CPAP mask modified with the application of silicon pads along the mask pillow cushion to optimize the CPAP mask-face model interface, primarily by adjustments to improve CPAP mask contact with the face model and limit the air leak during CPAP ventilation.

Once the patient's FDA-approved CPAP mask has been modified, the patient will then return to the BIDMC Specialties Clinic for a final fitting of the modified CPAP mask, with additional adjustments (as necessary) made to optimize the CPAP mask-patient interface. The study subject will then return home with his/her custom-modified CPAP mask to use as prescribed. Standard home monitoring and recording of use of the modified CPAP mask will be performed per usual case over a 30-day period. Data obtained during this 30-day period will focus on the duration of use of the modified CPAP mask, measurement of air leak and pressure loss, report of patient comfort and experience with the modified CPAP mask, and compare to data over a 30 day period using the CPAP mask prior to modification.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obstructive sleep apnea prescribed CPAP
* High air leak:1. Absolute high leak duration more than 15% of the use period and / or 2. Absolute high leak over 5% associated with periodic breathing.

Exclusion Criteria:

* Unable to wear full face CPAP
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Air leak time | 30 day
  Percent of air leak time over use of mask

SECONDARY OUTCOMES:
CPAP mask leak volume | 30 day
  Volume of leak recorded on CPAP machine
Epworth Sleepiness Scale | 30 day
  Sleepiness score - Likelihood of falling asleep in various daytime activities. Total Score Range 0-24.
Apnea Hypopnea Index | 30 day
  Apnea Hypopnea Index (events/hour)
CPAP Inspiratory pressure | 30 day
  Inspiratory pressure setting on CPAP machine (cm H2O)

CONTACTS AND LOCATIONS:
Overall Officials: Chee ChunMin, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States